CLINICAL TRIAL: NCT02474537
Title: An Open Label, Single-dose, Multi-center, Parallel-group, Two-staged Study to Evaluate Pharmacokinetics of Oral cMET Inhibitor INC280 in Non-Cancer Subjects With Impaired Hepatic Function and Non-Cancer Subjects With Normal Hepatic Function
Brief Title: INC280 in Healthy Subjects With Impaired Hepatic Function and Subjects With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINC280A2106
Record Dates: First submitted 2015-06-09; First posted 2015-06-17 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2019-03

CONDITIONS: Hepatic Impairment
Keywords: hepatic impairment,; INC280,; Oral cMET Inhibitor,; Non-Cancer
MeSH Terms: interventions — capmatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Normal hepatic function (Experimental): Subjects with normal hepatic function
  Interventions: Drug: INC280
- Mild hepatic impairment (Experimental): Subjects with mild hepatic impairment
  Interventions: Drug: INC280
- Moderate hepatic impairment (Experimental): Subjects with moderate hepatic impairment
  Interventions: Drug: INC280
- Severe hepatic impairment (Experimental): Subjects with severe hepatic impairment
  Interventions: Drug: INC280

INTERVENTIONS:
Drug: INC280 — Single 200 mg dose INC280

SUMMARY:
This is a phase I, multi-center, open-label, single oral dose, parallel group study to evaluate the pharmacokinetics and safety of INC280 in non-cancer subjects with impaired hepatic function and non-cancer subjects with normal hepatic function.The study population will be healthy male and postmenopausal or sterile female subjects who meet all of the inclusion and none of the exclusion criteria. Subjects will be assigned to groups according to their hepatic function: normal (Group 1), mild (Group 2), moderate (Group 3), and severe (Group 4) impairment. This study consists of a two-staged design with interim analysis. In Stage 1, subjects in Groups 1, 2 and 3 will be enrolled. Upon completion of Stage 1, an interim analysis will be conducted. Depending on the results of the analysis, either the study will conclude with no further enrollment or Stage 2 will commence with enrollment of Group 4.

A minimum of 6 evaluable subjects per group will be enrolled.Once enrolled in the study, participants will be confined to the facility for 4 days, given a single dose of INC280 and monitored for pharmacokinetic and safety assessments.

ELIGIBILITY:
Inclusion Criteria (all groups):

* Female subjects must be postmenopausal or sterile
* Good health, as determined by absence of clinically significant findings in medical history, physical examination, vital signs, and ECGs, unless it is consistent with known clinical disease for hepatic impairment subjects
* Adequate organ function and normal laboratory tests, unless it is consistent with known clinical disease for hepatic impairment subjects
* Body Mass Index (BMI) of 18- 36 kg/m2, with body weight ≥ 50 kg

Inclusion Criteria (hepatic impairment groups):

* Confirmed liver disease
* Stable comorbidities are allowed as long as generally considered healthy
* Subjects with hepatic impairment must meet the following laboratory values:
* Aspartate transaminase (AST) ≤ 5 x ULN
* Alanine transaminase (ALT) ≤ 5 x ULN
* Total bilirubin ≤ 3 x ULN (≤ 5 x XULN for subjects with severe hepatic impairment [group 4])
* Calculated creatinine clearance (using Cockcroft-Gault formula) ≥ 45 mL/min
* Platelets > 50 x 10^9/L. Subjects with severe hepatic impairment can be enrolled if platelet count > 40 x 10^9/L

Exclusion Criteria (all groups):

* History or presence of clinically significant ECG abnormalities or clinically significant cardiovascular disease
* Immunocompromised subjects, including HIV
* Use of drugs known to affect CYP3A4
* Use of QT-prolonging drugs
* Use of any other drugs, unless they are required to treat the hepatic impairment subject's disease
* Use of proton pump inhibitors (PPI) medications within 7 days prior to dosing and during the current study until last day of confinement

Exclusion Criteria (normal hepatic function group):

* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result

Exclusion Criteria (hepatic impairment groups):

* Active Grade 3 or 4 hepatic encephalopathy within 4 weeks of study entry
* Clinical evidence of severe ascites
* Ascites requiring paracentesis within 3 weeks prior to dosing

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-06-12 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-09-12 (Actual)

PRIMARY OUTCOMES:
AUClast of INC280 | Up to 72 hours post-dose
  INC280 pharmacokinetic parameters
AUCinf of INC280 | Up to 72 hours post-dose
  INC280 pharmacokinetic parameters
Cmax of INC280 | Up to 72 hours post-dose
  INC280 pharmacokinetic parameters
Tmax of INC280 | Up to 72 hours post-dose
  INC280 pharmacokinetic parameters
T1/2 of INC280 | Up to 72 hours post-dose
  INC280 pharmacokinetic parameters
CL/F of INC280 | Up to 72 hours post-dose
  INC280 pharmacokinetic parameters
Vz/F of INC280 | Up to 72 hours post-dose
  INC280 pharmacokinetic parameters

SECONDARY OUTCOMES:
Adverse events based on the CTCAE v4.03 grade (severity) and frequency, and other safety data (e.g., ECG, laboratory results) | Up to 30 days
  Safety
Unbound fraction and AUClast based on unbound concentration in plasma | 3 hours post-dose
  To assess the plasma protein binding of INC280
Unbound fraction and AUCinf based on unbound concentration in plasma | 3 hours post-dose
  To assess the plasma protein binding of INC280
Unbound fraction and Cmax based on unbound concentration in plasma | 3 hours post-dose
  To assess the plasma protein binding of INC280
Unbound fraction and Tmax based on unbound concentration in plasma | 3 hours post-dose
  To assess the plasma protein binding of INC280
Unbound fraction and T1/2 based on unbound concentration in plasma | 3 hours post-dose
  To assess the plasma protein binding of INC280
Unbound fraction and CL/F based on unbound concentration in plasma | 3 hours post-dose
  To assess the plasma protein binding of INC280
Unbound fraction and Vz/F based on unbound concentration in plasma | 3 hours post-dose
  To assess the plasma protein binding of INC280

CONTACTS AND LOCATIONS:
Overall Officials: NovartisPharmaceuticals, Study Director — NovartisPharmaceuticals
Locations (5):
- United States (5):
  - University of Miami Miller School of Medicine Clinical Resea Oncology, Miami, Florida
  - Clinical Pharmacology of Miami, LLC., Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota
  - Duke University Medical Center Oncology, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen X, Cui X, Pognan N, Quinlan M, Kapoor S, Rahmanzadeh G, Giovannini M, Marbury TC. Pharmacokinetics of capmatinib in participants with hepatic impairment: A phase 1, open-label, single-dose, parallel-group study. Br J Clin Pharmacol. 2022 Jan;88(1):91-102. doi: 10.1111/bcp.14929. Epub 2021 Jun 18. PMID 34046915
- See also: Results for CINC280A2106 can be found on the Novartis Clinical Trial Results website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17140